CLINICAL TRIAL: NCT00499083
Title: Neoadjuvant Intratumoral Injection of Dendritic Cells in Breast Cancer Translation of Biotechnology Into the Clinic
Brief Title: Paclitaxel, Cyclophosphamide & Doxorubicin, Autologous Dendritic Cells & Surgery in Stage II/III Breast Cancer (Women)
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University of Nebraska (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 0072-06-FB; P30CA036727 (NIH)
Record Dates: First submitted 2007-07-10; First posted 2007-07-11 (Estimated); Results first posted 2018-07-02 (Actual); Last update posted 2023-09-29 (Actual); Status verified 2023-09

CONDITIONS: Breast Cancer
Keywords: stage II breast cancer; stage IIIA breast cancer; stage IIIB breast cancer; stage IIIC breast cancer
MeSH Terms: conditions — Breast Neoplasms | interventions — Aromatase Inhibitors; Cyclophosphamide; Doxorubicin; liposomal doxorubicin; Paclitaxel; Albumin-Bound Paclitaxel; Tamoxifen; Gene Expression Profiling; Reverse Transcriptase Polymerase Chain Reaction; Immunoenzyme Techniques; Immunohistochemistry; Chemotherapy, Adjuvant; Biopsy; Neoadjuvant Therapy; Radiotherapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Vaccine (Experimental): Patients with HER-2/neu negative tumors will receive IT DCs one week after the first three of four cycles of dose dense T therapy and then four cycles of dose dense AC therapy will be given (i.e. T-AC).
  Interventions: Biological: therapeutic autologous dendritic cells; Drug: aromatase inhibition therapy; Drug: cyclophosphamide; Drug: doxorubicin hydrochloride; Drug: paclitaxel; Drug: tamoxifen citrate; Genetic: gene expression analysis; Genetic: protein expression analysis; Genetic: reverse transcriptase-polymerase chain reaction; Other: immunoenzyme technique; Other: immunohistochemistry staining method; Other: laboratory biomarker analysis; Procedure: adjuvant therapy; Procedure: biopsy; Procedure: conventional surgery; Procedure: neoadjuvant therapy; Radiation: radiation therapy

INTERVENTIONS:
Biological: therapeutic autologous dendritic cells — injected into the primary breast mass or palpable axillary node, one week after the first, second and third T treatments. If, after a cycle(s) of chemotherapy, no tumor can be localized by ultrasound, the DCs will be injected where the tumor bed was localized by the clip or marker.
Drug: aromatase inhibition therapy — Adjuvant hormone therapy for patients having tumors with estrogen and/or progesterone receptors. Premenopausal patients will be treated with tamoxifen. Post or perimenopausal women may receive tamoxifen or an aromatase inhibitor (AI) or those drugs in sequence as determined by the treating oncologist. Hormone therapy will be given for at least 5 years.
  Other Names: endocrine therapy
Drug: cyclophosphamide — 600 mg/m2 IV day 1 every 2 weeks for 4 cycles
  Other Names: Cytoxan
Drug: doxorubicin hydrochloride — 60 mg/m2 IV day 1 every 2 weeks for 4 cycles
  Other Names: Lipodox, Lipodox 50, and Doxil
Drug: paclitaxel — 175 mg/m2 intravenously (IV) over at least 3 hours day 1 every 2 weeks for 4 cycles.
  Other Names: Abraxane
Drug: tamoxifen citrate — Adjuvant hormone therapy for patients having tumors with estrogen and/or progesterone receptors. Premenopausal patients will be treated with tamoxifen. Post or perimenopausal women may receive tamoxifen or an aromatase inhibitor (AI) or those drugs in sequence as determined by the treating oncologist. Hormone therapy will be given for at least 5 years.
  Other Names: Nolvadex
Genetic: gene expression analysis — IHC for CEA and Survivin with appropriate controls will be done on the tumor biopsy material (preferably from the initial diagnostic biopsy).
Genetic: protein expression analysis — Tumor biopsymaterial (preferably from the initial diagnostic biopsy) will be stained by IHC with appropriate controls for COX-2, VEGF A, T cell and Dendritic Cell infiltration.
Genetic: reverse transcriptase-polymerase chain reaction — delta Ct (quantitative real time- reverse transcription-polymerase chain reaction (qRT-PCR)) of COX-2 and VEGF will be divided into the upper or lower median and Fisher Exact test used to assess the difference in response.
Other: immunoenzyme technique — Estrogen and progesterone receptor, Her2/neu testing: Tumor biopsy material (preferably the initial diagnostic biopsy if tissue is available) will be examined by Immunohistochemistry (IHC) with appropriate controls for estrogen, progesterone receptors and Her2/neu. If the IHC is 2+ or in the indeterminate range, further testing of over-expression of Her2/neu by fluorescent in situ hybridization (FISH) will be done . If this has already been done and reported by the referring hospital, it will not be repeated. These tests are standard of care.
  CEA and Survivin testing: IHC for CEA and Survivin with appropriate controls will be done on the tumor biopsy material (preferably from the initial diagnostic biopsy).
  COX-2 and VEGF A , T cell and Dendritic Cells: Tumor biopsymaterial (preferably from the initial diagnostic biopsy) will be stained by IHC with appropriate controls for COX-2, VEGF A, T cell and Dendritic Cell infiltration.
Other: immunohistochemistry staining method — Estrogen and progesterone receptor, Her2/neu testing: Tumor biopsy material (preferably the initial diagnostic biopsy if tissue is available) will be examined by Immunohistochemistry (IHC) with appropriate controls for estrogen, progesterone receptors and Her2/neu. If the IHC is 2+ or in the indeterminate range, further testing of over-expression of Her2/neu by fluorescent in situ hybridization (FISH) will be done . If this has already been done and reported by the referring hospital, it will not be repeated. These tests are standard of care.
  CEA and Survivin testing: IHC for CEA and Survivin with appropriate controls will be done on the tumor biopsy material (preferably from the initial diagnostic biopsy).
  COX-2 and VEGF A , T cell and Dendritic Cells: Tumor biopsymaterial (preferably from the initial diagnostic biopsy) will be stained by IHC with appropriate controls for COX-2, VEGF A, T cell and Dendritic Cell infiltration.
Other: laboratory biomarker analysis — Estrogen and progesterone receptor, Her2/neu testing: Tumor biopsy material (preferably the initial diagnostic biopsy if tissue is available) will be examined by Immunohistochemistry (IHC) with appropriate controls for estrogen, progesterone receptors and Her2/neu. If the IHC is 2+ or in the indeterminate range, further testing of over-expression of Her2/neu by fluorescent in situ hybridization (FISH) will be done . If this has already been done and reported by the referring hospital, it will not be repeated. These tests are standard of care.
  CEA and Survivin testing: IHC for CEA and Survivin with appropriate controls will be done on the tumor biopsy material (preferably from the initial diagnostic biopsy).
  COX-2 and VEGF A , T cell and Dendritic Cells: Tumor biopsymaterial (preferably from the initial diagnostic biopsy) will be stained by IHC with appropriate controls for COX-2, VEGF A, T cell and Dendritic Cell infiltration.
Procedure: adjuvant therapy — Hormone manipulation Adjuvant hormone therapy for patients having tumors with estrogen and/or progesterone receptors. Premenopausal patients will be treated with tamoxifen. Post or perimenopausal women may receive tamoxifen or an aromatase inhibitor (AI) or those drugs in sequence as determined by the treating oncologist. Hormone therapy will be given for at least 5 years.
Procedure: biopsy — Two tumor biopsies will be performed. The first tumor biopsy will be performed before apheresis for diagnostic purposes, and again after completion of the first four chemotherapy treatments. Patients will undergo local anesthesia with lidocaine and 1% epinephrine followed by 1-2 core biopsies of the breast primary and/or palpable axillary node with a 14 gauge, 16 cm. Bard needle or other similar needle. The procedure may be done under ultrasound guidance. If a metal clip or marker has not been previously placed in the tumor, it will be placed before treatment.
Procedure: conventional surgery — Definitive breast surgery Surgery will occur two to four weeks after the last course of chemotherapy. Modified radical mastectomy or lumpectomy and standard axillary dissection could be performed and the specific procedure will be decided by the patient and physician team. If a sentinel node dissection was done prior to chemotherapy and was negative, no further node dissection is necessary. A standard node dissection will be necessary if no node assessment was done prior to chemotherapy or if the pre- chemotherapy sentinel node was positive.
Procedure: neoadjuvant therapy — Chemotherapy: Paclitaxel (T) 175 mg/m2 intravenously (IV) over at least 3 hours day 1. Repeat every 2 weeks for 4 cycles. IT DCs will be injected into the primary breast mass or palpable axillary node, one week after the first, second and third T treatments.
Radiation: radiation therapy — Radiation therapy Radiation is started two to four weeks after surgery for all patients receiving lumpectomy and those patients after mastectomy that the physician feels chest wall radiation is warranted (example: T3 or T4 breast lesion, four or more axillary nodes etc.). The exact doses and methods of administration will be determined by the treating radiation therapist, but should be standard breast radiotherapy and not partial breast or investigational methods.

SUMMARY:
RATIONALE: Drugs used in chemotherapy, such as paclitaxel, cyclophosphamide, and doxorubicin, work in different ways to stop the growth of tumor cells, either by killing the cells or by stopping them from dividing. Injecting the patient's dendritic cells directly into the tumor may stimulate the immune system and stop tumor cells from growing. Radiation therapy uses high-energy x-rays to kill tumor cells. Estrogen can cause the growth of breast cancer cells. Hormone therapy using tamoxifen may fight breast cancer by blocking the use of estrogen by the tumor cells. Giving combination chemotherapy together with autologous dendritic cells before surgery may make the tumor smaller and reduce the amount of normal tissue that needs to be removed. Giving radiation therapy and hormone therapy after surgery may kill any tumor cells that remain after surgery.

PURPOSE: This phase II trial is studying the side effects and how well giving paclitaxel together with cyclophosphamide and doxorubicin followed by autologous dendritic cells and surgery with or without radiation therapy and/or hormone therapy works in treating women with stage II or stage III breast cancer.

DETAILED DESCRIPTION:
OBJECTIVES:

* Assess the safety of intratumoral (IT) autologous dendritic cell (DC) injection in women with stage II or III breast cancer receiving neoadjuvant paclitaxel, cyclophosphamide, and doxorubicin hydrochloride followed by surgery with or without adjuvant radiotherapy and/or hormone therapy.
* Determine the clinical and pathologic response in patients treated with this regimen.
* Determine the immune response, in terms of tumor cell apoptosis and the presence and characterization of tumor infiltrating white blood cells in resected breast cancer, in patients treated with this regimen.
* Determine if IT DC injections administered during neoadjuvant chemotherapy-induced tumor cell apoptosis can induce T-cell responses to tumor antigens in these patients.

OUTLINE: This is an open-label study.

* Leukapheresis: Patients undergo leukapheresis at baseline to collect peripheral blood mononuclear cells for dendritic cell (DC) culture.
* Neoadjuvant, dose-dense chemotherapy: Patients receive paclitaxel IV over at least 3 hours on day 1 and filgrastim (G-CSF) subcutaneously (SC) on days 4-14 or pegfilgrastim SC on day 2. Treatment repeats every 2 weeks for up to 4 courses in the absence of disease progression or unacceptable toxicity.

Beginning 2 weeks after completion of paclitaxel chemotherapy, patients receive cyclophosphamide IV and doxorubicin hydrochloride IV on day 1 and G-CSF SC on days 4-14 or pegfilgrastim SC on day 2. Treatment repeats every 2 weeks for up to 4 courses in the absence of disease progression or unacceptable toxicity.

* Intratumoral injection of autologous DCs: Intratumoral autologous DCs are injected into the primary breast mass or palpable axillary node on day 7 of the 1st, 2nd, and 3rd courses of paclitaxel chemotherapy. If no tumor can be localized by ultrasound after a course of chemotherapy, the DCs are then injected into the site of the tumor bed previously localized by clip or marker. In the event that the previously injected primary tumor cannot be localized by ultrasound, a palpable lymph node, if still present, should be injected rather than the tissue next to the primary tumor clip or marker.
* Definitive breast surgery: Within 2-4 weeks after completion of neoadjuvant chemotherapy, patients undergo modified radical mastectomy or lumpectomy with or without standard axillary node dissection.* NOTE: *Standard axillary node dissection is only required if no node assessment was done prior to chemotherapy or if the pre-chemotherapy sentinel node was positive.
* Radiotherapy: Patients undergoing lumpectomy or those with residual disease requiring chest wall radiotherapy after mastectomy (e.g., T3 or T4 breast lesions or 4 or more axillary lymph nodes) undergo radiotherapy 2-4 weeks after surgery.
* Hormone therapy: Patients with estrogen and/or progesterone receptor-positive tumors receive adjuvant hormone therapy for ≥ 5 years. Premenopausal patients receive tamoxifen citrate and post- or perimenopausal patients receive either tamoxifen citrate or an aromatase inhibitor (AI), or both of these drugs in sequence, as determined by the treating oncologist.

Peripheral blood samples are obtained during each DC injection, at staging/biopsy, and then periodically for up to 2 years. Blood samples are analyzed by ELISPOT and ELISA assays for evaluation of immune response.

Tumor tissue is obtained by core biopsy of the breast primary and/or palpable axillary lymph node at baseline and again after completion of paclitaxel chemotherapy. Tumor tissue is analyzed by IHC and RT-PCR for COX-2 and VEGF-A and -C expression levels, as well as T-cell and DC infiltration of the tumor. T-cell and DC infiltration is evaluated for correlation with clinical outcomes at diagnosis, at the midpoint biopsy following paclitaxel chemotherapy, and at definitive surgery.

After completion of study therapy, patients are followed periodically for up to 2 years.

ELIGIBILITY:
Inclusion Criteria:

* Histologically confirmed invasive breast cancer meeting the following criteria:

  * Primary tumor ≥ 3 cm by mammography, ultrasound, or palpation AND/OR palpable axillary lymph nodes > 1 cm
  * Survivin- and/or carcinoembryonic antigen-positive by IHC
  * Tumor must be localized by exam or ultrasound to allow tumor injection
  * No stage IV or metastatic disease
* HER2/neu-negative tumor by IHC

  o If 2+ or in the indeterminate range, further testing of HER2/neu overexpression by fluorescent in situ hybridization (FISH) is required
* Hormone receptor status known
* Female
* Pre-, peri-, or postmenopausal
* ECOG performance status 0-1
* Fertile patients must use effective contraception during and for up to 6 months following completion of study therapy
* ANC ≥ 1,500/mm³
* Platelet count ≥ 100,000/mm³
* Alkaline phosphatase ≤ 1.5 times upper limit of normal (ULN)
* Total bilirubin ≤ 1.5 times ULN
* AST and ALT ≤ 1.5 times ULN
* Creatinine < 1.5 times ULN

Exclusion Criteria:

* No prior chemotherapy or radiotherapy
* No active serious infections
* No prior malignancy except adequately treated basal cell or squamous cell skin cancer, noninvasive carcinoma, or other cancer from which the patient has been disease free for 5 years
* No comorbidity or condition that would interfere with study assessments and procedures or preclude study participation
* Not pregnant or nursing/negative pregnancy test

Ages: 19 Years to 120 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 17 (Actual)
Dates: Start 2006-05-01 (Actual); Primary Completion 2009-07-01 (Actual); Study Completion 2010-01-28 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Elizabeth C Reed, MD, Principal Investigator — University of Nebraska; Kenneth H Cowan, MD, PhD, Principal Investigator — University of Nebraska
Locations (2):
- United States (2):
  - H. Lee Moffitt Cancer Center and Research Institute, University of South Florida, Tampa, Florida
  - Eppley Cancer Center, University of Nebraska Medical Center, Omaha, Nebraska

REFERENCES:
- [Derived] Hong WX, Sagiv-Barfi I, Czerwinski DK, Sallets A, Levy R. Neoadjuvant Intratumoral Immunotherapy with TLR9 Activation and Anti-OX40 Antibody Eradicates Metastatic Cancer. Cancer Res. 2022 Apr 1;82(7):1396-1408. doi: 10.1158/0008-5472.CAN-21-1382. PMID 35135810

RESULTS

PARTICIPANT FLOW:
Groups:
- Vaccine: Patients with HER-2/neu negative tumors received therapeutic autologous dendritic cells: injected into the primary breast mass or palpable axillary node, one week after the first, second and third T treatments.
  Adjuvant hormone therapy for patients having tumors with estrogen and/or progesterone receptors. Premenopausal patients will be treated with tamoxifen. Post or perimenopausal women may receive tamoxifen or an aromatase inhibitor.
  Patients received 4 cycles of paclitaxel: 175 mg/m2 (IV), followed by 4 cycles of cyclophosphamide: 600 mg/m2 IV and doxorubicin hydrochloride: 60 mg/m2 IV in a bi-weekly dose dense fashion
  All patients had pre-treatment biopsy and second tumor biopsy after 4 cycles of paclitaxel to evaluate responses to the dendritic cell injections.
Period: Overall Study
Arm/Group | Vaccine
Started | 17
Participants at UNMC | 3
Participants at Moffitt Cancer Center | 14
Completed | 14
Not Completed | 3
Not completed — Not evaluable | 3

BASELINE CHARACTERISTICS:
Population: Numbers are based on number of evaluable participants.
Arm/Group | Vaccine
Number analyzed (Participants) | 14
Age, Continuous [Median (Full Range); unit: years] | 51.5 [NA to NA] — Only median value available from existing documentation, no other documentation exists.
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 14
  Male | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 14

OUTCOME MEASURES:

1. Primary Outcome: Number of Patients With Pathological Complete Response
Description: Assessed by the institutional pathologist.
  * Grade 1: disappearance of all tumor on microscopic assessment in the breast and LNs
  * Grade 2: presence of in situ carcinoma only in the breast, no invasive tumor, and no tumor found in the LNs
  * Grade 3: presence of invasive carcinoma with stromal alteration, such as sclerosis or fibrosis
  * Grade 4: no or few modifications of the tumor appearance
Time Frame: At definitive surgery.
Measure: Number; unit: participants
Arm/Group | Vaccine
Number analyzed (Participants) | 14
participants | 2

2. Secondary Outcome: Inflammatory Cell Infiltration
Description: T cell response to tumor-specific Ag, will be measured by ELISPOT assay with a biologic response defined as double the average ELISPOT reactivity in post-vaccination peripheral blood (PB) compared to pre-vaccination PB.
Time Frame: Post-vaccination peripheral blood (PB) after the last chemotherapy.
Population: Evaluation of this data is unknown as was not provided by collaborating center performing the analysis.
Arm/Group | Vaccine
Number analyzed (Participants) | 0

3. Secondary Outcome: Antibody-dependent Cell-mediated Cytotoxicity
Description: as for outcome 2
Time Frame: Post-vaccination peripheral blood (PB) after the last chemotherapy.
Population: Evaluation of this data is unknown as was not provided by collaborating center performing the analysis.
Arm/Group | Vaccine
Number analyzed (Participants) | 0

4. Secondary Outcome: Influence of Tumor COX-2 and VEGF Expression on Dendritic Cell-mediated Tumor-specific Immunity
Description: as for outcome 2
Time Frame: Post-vaccination peripheral blood (PB) after the last chemotherapy.
Population: Evaluation of this data is unknown as was not provided by collaborating center performing the analysis.
Arm/Group | Vaccine
Number analyzed (Participants) | 0

ADVERSE EVENTS:
Time Frame: Adverse events were collected from the time of when patients consented to the study until 30 day after completion of the study treatment, up to 6 months.
Description: Grade 3/4 toxicities were collected for this study. Complete evaluation of this data is unknown. We only have adverse event data from UNMC.
Arm/Group | Vaccine
All-Cause Mortality (participants affected / at risk) | 0/3
Serious Adverse Events (participants affected / at risk) | 1/3
Other Adverse Events (participants affected / at risk) | 3/3
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Vaccine (N=3)
Febrile neutropenia (Blood and lymphatic system disorders) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Vaccine (N=3)
Thromboembolic event (Vascular disorders) | 1 (1)
hypokalemia (Metabolism and nutrition disorders) | 1 (1)
mucositis oral (Gastrointestinal disorders) | 1 (1)
palmar-plantar erythrodysesthesia (Skin and subcutaneous tissue disorders) | 1 (1)
bone pain (Musculoskeletal and connective tissue disorders) | 1 (1)
white blood cell decreased (Investigations) | 1 (1)
neutrophil count decreased (Investigations) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No